CLINICAL TRIAL: NCT06366503
Title: A Randomized, Single-Center, Double-Blinded, Split-Face, Controlled Study Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With Fractional Ablative CO2 Laser for Facial Rejuvenation
Brief Title: Evaluating Procedure Pairing of a Post-Procedure Cream Versus a Comparator in Patients Treated With Fractional Ablative CO2 Laser for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RS-2023-05
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-04

CONDITIONS: Photoaging; Wrinkle; Skin Laxity
Keywords: post-procedure; Fractional Ablative CO2 Laser
MeSH Terms: conditions — Cutis Laxa | interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Randomized, Single-Center, Double-Blinded, Split-Face, Controlled
Who Masked: Participant, Investigator
Masking Description: Subjects were randomly assigned to use the active post-procedure cream on one side of the face and the comparator anhydrous formulation on the opposite side of the face.
  The products were packaged in the same container and labelled post-procedure cream. This was a double blinded study, where the investigator, study subject, and other study personnel involved in the evaluation of the efficacy or safety were blinded to group during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Split-Face Application of Active (Experimental) (Experimental): Active (Experimental) Post-Procedure Cream
  Dosage Form: reverse emulsion (water in oil) cream containing bioactive ingredients, botanical actives, peptides, and antioxidants.
  Frequency of Dosage: Three times daily (morning, afternoon, and evening). Subjects were asked to apply face (including upper eyelid), jawline, and neck. The product was labelled with Right or Left depending on split-face randomization.
  Study duration: 28 days. Active Post-Procedure Cream duration 14-days.
  Interventions: Procedure: Fractional Ablative CO2 Laser; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen
- Split-Face Application of Comparator (Active Comparator): COMPARATOR:
  Dosage Form: anhydrous formulation.
  Comparator Anhydrous Formulation Frequency of Dosage: Three times daily (morning, afternoon, and evening). Subjects were asked to apply on the face (including upper eyelid), jawline, and neck. The product was labelled with Right or Left depending on split-face randomization.
  Study duration: 28 days. Comparator duration 14-days.
  Interventions: Procedure: Fractional Ablative CO2 Laser; Other: Facial Cleanser; Other: Facial Moisturizer; Other: Sunscreen; Other: Basic Ointment

INTERVENTIONS:
Procedure: Fractional Ablative CO2 Laser — A fractional ablative DEKA SmartXide Tetra CO2 laser treatment was performed after a 14-day washout period. Subjects were numbed for 1 hour prior to procedure with topical numbing cream (lidocaine 23%, tetracaine 7%). The global face was treated with a single pass. Treatment parameters include power 20 W, spacing 500 um (13% density), Dwell time 1200 us DEKA pulse mode, spray mode on.
  Other Names: DEKA SmartXide Tetra CO2 laser treatment
Other: Facial Cleanser — Facial cleanser was to be used by subjects twice daily during the 14-day washout period and three times daily during the 14-day post-procedure timeline.
  Other Names: Gentle Foaming Cleanser, Revision Skincare
Other: Facial Moisturizer — A bland facial moisturizer was to be used by subjects twice daily during the 14-day washout period and three times daily between day 3 and 14 post-procedure. Two pumps were to be applied to the face (avoiding the upper eyelid) after applying the active and comparator.
Other: Sunscreen — During the 14-day washout period, a bland sunscreen was to be used by subjects in the morning after cleansing and facial moisturizer application with reapplications as needed throughout the day per FDA recommendations. For days 3-14 post-procedure, the bland sunscreen was to be used daily by subjects in the morning and afternoon after cleansing, split-face application of the active post-procedure cream and comparator anhydrous formulation, and facial moisturizer application.
  Other Names: Neutrogena Sheer Zinc SPF 50
Other: Basic Ointment — The basic ointment was used only on the comparator side for three days (72 hours) post-procedure. This was a requirement of the comparator anhydrous formulation.
  Other Names: Vanicream Moisturizing Ointment
  Arms: Split-Face Application of Comparator

SUMMARY:
This randomized, single-center, double-blinded, split-face, controlled clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after fractional ablative CO2 laser treatment and for 14 days post-procedure with three times daily application in healthy female subjects aged 35 to 65 with moderate to severe global facial overall photodamage (score of 4 to 9 out of the 10-point Modified Griffiths' scale). Furthermore, this clinical trial compared the active post-procedure cream to a comparator anhydrous formulation often paired with skin rejuvenation procedures. This is a cosmetic study with a FDA-regulated device.

A total of 22 healthy female subjects completed the study.

DETAILED DESCRIPTION:
This randomized, single-center, double-blinded, split-face, controlled clinical trial was conducted to investigate the tolerability, safety, and efficacy of a post-procedure cream when used immediately after fractional ablative CO2 laser treatment and for 14 days post-procedure with three times daily application in healthy female subjects aged 35 to 65 with moderate to severe global facial overall photodamage (score of 4 to 9 out of the 10-point Modified Griffiths' scale). The ability of the post-procedure cream to soothe skin and improve patient downtime post-procedure was investigated by evaluating tolerability parameters (erythema, edema, dryness, burning, itching, stinging) and pain over the course of the study. Furthermore, this clinical trial compared the active post-procedure cream to a comparator anhydrous formulation often paired with skin rejuvenation procedures.

A 14-day washout period was required of all subjects prior to CO2 laser treatment. Tolerability (investigator: erythema, edema, dryness; subject: burning, itching, stinging) and safety were assessed through grading at screening, pre-procedure, post-procedure, post-procedure/post-product application, and days 1, 3, 5, 7, and 14 post-procedure. Pain evaluations were completed by subjects using the 11-point Wong Baker Faces® Pain Rating scale post-procedure, post-procedure/post-product application, and days 1, 3, 5, 7, and 14 post-procedure.

In addition, efficacy evaluation using the Modified Griffiths' scale was performed at screening, pre-procedure, and days 1, 3, 5, 7, and 14 post-procedure. Self-assessment questionnaires were completed by subjects post-procedure/post-product application and days 1, 3, and 14 post-procedure. Clinical photography was completed at all timepoints (screening to day 14 post-procedure).

A total of 22 subjects completed study participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects 35-65 years of age
* Fitzpatrick Skin Type I to III
* Any race or ethnicity
* Moderate to Severe Overall Photodamage (global face) (score of 4 to 9 out of the 10-point Modified Griffiths' scale, where 0 = none and 9 = severe)
* No known medical conditions that, in the Investigator's opinion, may interfere with study participation.
* Willing to discontinue all active topical facial products and only use the assigned test products for the duration of the study.
* Female subjects of childbearing potential must be willing to use a form of birth control during the study.

Exclusion Criteria:

* Nursing, pregnant, or planning a pregnancy during this study.
* Having undergone a chemical peel, microdermabrasion, hydro dermabrasion or anti-aging facial within 1 month; non-ablative laser (including IPL) or non-ablative fractional laser resurfacing of the face within 6 months; ablative laser resurfacing of the face within 12 months.
* Not willing to discontinue active topical facial products for 14 days prior to the Baseline Visit

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Investigator Tolerability | 14 days
  The primary tolerability endpoint will be Investigator Tolerability Assessment of erythema, edema, and dryness. A change in score or lack of significant change post product application, Day 1 (24 hours), Day 3, Day 5, Day 7, and Day 14 in comparison to baseline (immediately post-procedure) indicates tolerability / safety of the test material.
  A four-point scale will be used with a lower score indicating a better outcome:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
Incidence of Adverse Events | 14-days
  The primary safety endpoint will be determined by the incidence and severity of adverse events in healthy subjects, including immediately post-procedure and throughout the length of the study.
Subject Tolerability | 14 days
  The subject tolerability endpoint will be Subject Tolerability Assessment of burning, itching, and stinging. A change in score or lack of significant change post product application, Day 1 (24 hours), Day 3, Day 5, Day 7, and Day 14 in comparison to baseline (immediately post-procedure) indicates tolerability / safety of the test material.
  A four-point scale will be used with a lower score indicating a better outcome:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe

SECONDARY OUTCOMES:
Self-Assessment Questionnaire | 14 days
  A change in response values at Day 1 (24 hours), Day 3, and Day 14 compared to post-procedure/post-product application response values indicates an improvement. Baseline responses will be set to post-procedure/post-product application. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement / question being asked.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Weir, MD, PhD, Principal Investigator — The Dermatology Group
Locations (1):
- The Dermatology Group, Blue Ash, Ohio, United States

REFERENCES:
- [Derived] Weir NM, Burns AJ, Kononov T, Zahr AS. A Novel Neurocosmetic Postprocedure Cream for Optimal Recovery and Tolerability From Energy-Based Devices. Lasers Surg Med. 2025 Dec;57(10):788-798. doi: 10.1002/lsm.70078. Epub 2025 Nov 24. PMID 41286587